CLINICAL TRIAL: NCT01632033
Title: Estimation de la capacité Fonctionnelle a la Marche Par Questionnaire Clinique Chez Des Patients adressés Pour Bilan artériel Des Membres inférieurs: Etude WELCH-bis
Brief Title: Functional Evaluation With Questionnaire in Patients Investigated for Suspected Peripheral Artery Disease
Acronym: WELCH-bis
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PL 2012/14
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral artery disease; claudication; walking; questionnaire
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Investigation for lower limb arteries: Patients referred for investigation of assumed peripheral artery disease (PAD)

SUMMARY:
The purpose of this study is to test the routine faisibility of a questionnaire to estimate walking impairment(The WELCH questionnaire) in patients investigated for suspected PAD.

DETAILED DESCRIPTION:
The WELCH and WIQ questionnaires are self completed by the patients and scored by the physician after self-completion.

ELIGIBILITY:
Inclusion Criteria:

* Sigjned consent for the data treatment as a database

Exclusion Criteria:

* Non french native language age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for arterial leower limb investigations
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Scoring of the WELCH. Percent scored questionnaires | 1 day
  Predetermined scored . Scoring is optional and compared to scoring of the WIQ

CONTACTS AND LOCATIONS:
Overall Officials: Denise JOLIVOT, MD, Study Chair — University Hospital, Angers
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Ouedraogo N, Chanut M, Aubourg M, Le Hello C, Hidden V, Audat G, Harbonnier M, Abraham P. Development and evaluation of the Walking Estimated-Limitation Calculated by History questionnaire in patients with claudication. J Vasc Surg. 2013 Oct;58(4):981-8. doi: 10.1016/j.jvs.2013.03.039. Epub 2013 May 7. PMID 23663870